CLINICAL TRIAL: NCT00518362
Title: To Compare the Efficacy and Safety of TW vs Valsartan in the DN
Brief Title: To Compare the Efficacy and Safety of Tripterygium (TW) Versus Valsartan in the Diabetic Nephropathy (DN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-0701
Record Dates: First submitted 2007-08-16; First posted 2007-08-20 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-04

CONDITIONS: Diabetic Nephropathy
Keywords: TW; Valsartan; treatment; diabetic nephropathy; Proteinuria
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- immunosuppressor (Experimental): Valsartan,160mg/d,TW 120mg/d
  Interventions: Drug: TW

INTERVENTIONS:
Drug: TW — TW,120 mg/d

SUMMARY:
The purpose of this study is to compare the efficacy and safety of Tripterygium (TW) versus Valsartan (ARB) in the Diabetic Nephropathy (DN).

DETAILED DESCRIPTION:
Diabetic nephropathy with heavy proteinuria have high risks of progressing to end stage renal disease. Though recent studies have shown that ACEI or ARB could reduce proteinuria of DN and slowed the progression to ESRD. But ARBs can only reduce proteinuria about 30%, so some patients still have heavy proteinuria,and then loss their renal function rapidly. So, to reduce the proteinuria of DN is a very important therapy target.

Tripterygium (TW) is a Chinese traditional patent drug, it can reduce proteinuria of chronic glomerular nephritis. So, we designed this randomized, prospective clinical trial to assess the efficacy and safety of TW versus ARB in the treatment of heavy proteinuria of DN.

ELIGIBILITY:
Inclusion Criteria:

1. A new diagnosis of diabetic nephropathy proved by histology and(or) serology.
2. Proteinuria > 2.5 g/24 h
3. serum creatinine < 3 mg/dl
4. age 35-65 years

Exclusion Criteria:

1. Co-existence of anther chronic glomerular nephritis.
2. Severe disfunction of the liver
3. White blood cell < 3000/ul
4. Severe infection in the past 1 month
5. Malignant hypertension which in hard to control
6. Myocardial infarct or heart failure or sever cerebral vessels complication in the past 6 month

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To access the efficacy of TW compared to ARB in treatment of heavy proteinuria of diabetic nephropathy | 6 months

SECONDARY OUTCOMES:
To investigate the safety and tolerability of TW vs ARB. To access whether TW can delay the progression to ESRD or creatinine-doubling in diabetic nephropathy with heavy proteinuria. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, Master, Principal Investigator — Jinling Hospital, China
Locations (1):
- Research Institute of Nephrology, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Ge Y, Xie H, Li S, Jin B, Hou J, Zhang H, Shi M, Liu Z. Treatment of diabetic nephropathy with Tripterygium wilfordii Hook F extract: a prospective, randomized, controlled clinical trial. J Transl Med. 2013 May 31;11:134. doi: 10.1186/1479-5876-11-134. PMID 23725518